CLINICAL TRIAL: NCT07025135
Title: Evaluation of the Effectiveness of a Mobile Application in the Treatment of Children With Functional Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NKBBN/920/2021
Record Dates: First submitted 2025-05-30; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Constipation - Functional
Keywords: functional constipation; pediatrics; mobile app

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient-caregiver dyad using mobile app (Experimental): Patient-caregiver dyad receives standard care (optimal macrogol treatment) plus access to dedicated mobile app
  Interventions: Behavioral: comparison between use of mobile app
- patient-caregiver dyad using paper recommendation (Active Comparator): Patient-caregiver dyad receives standard care (optimal macrogol treatment) plus a non-interactive, educational-only printed version of recommendations.
  Interventions: Behavioral: Patient-caregiver dyad using printed recommendations

INTERVENTIONS:
Behavioral: comparison between use of mobile app — Patient-caregiver dyad receive standard care (optimal macrogol treatment) plus a mobile app featuring symptom tracking, medication reminders, dietary tips, and gamification elements.
  Arms: patient-caregiver dyad using mobile app
Behavioral: Patient-caregiver dyad using printed recommendations — Patient-caregiver dyad receives standard care ( optimal macrogol treatment) plus a non-interactive, educational-only printed version of recommendations.
  Arms: patient-caregiver dyad using paper recommendation

SUMMARY:
This randomized, double-blind clinical trial evaluates the effectiveness of use of a mobile health application in supporting the treatment of functional constipation in children aged 4 to 18 years. Participants are randomly assigned ( with en-bloc randomization) to either an intervention group using an interactive app with symptom tracking, reminders, and games or a control group using equivalent, but printed materials. The primary outcome is the improvement in constipation symptoms after 3 months with follow-up after 6 months (+/- 30 days) after enrollment. Secondary outcomes include achieving regular bowel movements. The study aims to determine whether digital tools can enhance treatment adherence and clinical outcomes in pediatric functional constipation.

DETAILED DESCRIPTION:
Functional constipation is a common pediatric disorder that significantly affects the quality of life of children and their families. Despite the availability of evidence-based guidelines such as the Rome IV criteria and the ESPGHAN/NASPGHAN (European Society for Paediatric Gastroenterology, Hepatology and Nutrition/ North American Society for Paediatric Gastroenterology, Hepatology and Nutrition recommendations, treatment adherence remains a major challenge, often leading to suboptimal outcomes and chronic symptoms.

This randomized, double-blind, parallel-group clinical trial investigates the efficacy of a mobile health application designed to support the treatment of functional constipation in children. The study is conducted among children aged 4 to 18 years who meet the Rome IV diagnostic criteria for functional constipation. Participants are randomly allocated in a 1:1 ratio into two groups: an intervention group receiving standard care supplemented with an interactive mobile app, and a control group receiving standard care with a printed version of recommendations.

The interactive mobile app includes features aimed at increasing engagement and adherence, such as daily symptom tracking, medication and hydration reminders, educational content, diet guidance, and rewards to motivate participation. The printed materials are equivalent to app regarding information.

This trial aims to determine whether a digital intervention can meaningfully enhance treatment adherence and improve clinical outcomes in pediatric functional constipation, and potentially serve as a scalable tool for supporting families in managing this common chronic condition.

The primary endpoint is the improvement in constipation symptoms over 3 months and 6 months follow-up, assessed by measuring quality of life (measured using the PedsQL Gastrointestinal Module). Secondary outcome is the improvement (bowel movement frequency and stool consistency using the Bristol Stool Form Scale).

Data collection: Symptoms tracking - PedsQL Gastrointestinal Module, bowel movements, water intake, macrogol intake

*Mobile App Features:

Daily symptom tracking

Medication reminders

Diet and fluid intake tips

Games and reward system

Control: Identical interface without interactive features

Intervention scheme:

Visit 1 (enrolment, 0):

medical history, physical examination interpretation of laboratory findings (coeliac disease, vitamin D deficiency, hypercalcemia, hypothyroidism), which would exclude patient from study app presentation or printed materials introduction PedsQL Gastrointestinal Module fill-up

Visit 2 (after 1 month, 1)

medical history, physical examination counseling PedsQL Gastrointestinal Module fill-up and comparison of results from previous visit

Visit 3 (after another 1 month, 2)

medical history, physical examination PedsQL Gastrointestinal Module fill-up and comparison of results from previous visit

Visit 4 (after another 1 month, 3)

medical history, physical examination counseling PedsQL Gastrointestinal Module fill-up and comparison of results from previous visit

Visit 5 ( follow-up after 6 month of study, 6) medical history, physical examination counseling, program ending and final remarks PedsQL Gastrointestinal Module fill-up and comparison of results from previous visit

ELIGIBILITY:
Inclusion Criteria:

* age 4-18,
* meeting Rome Criteria IV of functional constipation

Exclusion Criteria:

* organic causes of constipation
* comorbidities

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
improvement of symptoms | 6 month +/- 30 days
  Decreased severity (measured by Likert scale, where 0 means never and 5 means almost always) of symptoms measured by PedsQL (Pediatric Quality of Life) - Gastrointestinal Module

SECONDARY OUTCOMES:
Achieving regularity of bowel movements | 6 months +/-30 days
  Number of participants with regular bowel movement (more than 2 bowel movements/week)

CONTACTS AND LOCATIONS:
Locations (1):
- Department and Clinic of Pediatrics, Gastroenterology, Allergology and Pediatric Nutrition of Medical University of Gdansk, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
anyone contacting the authors will be assessed and data will be given to researchers/public authorities
Supporting Information: Study Protocol, ICF, CSR
Access Criteria: anyone contacting the authors will be assessed and data will be given to researchers/public authorities

REFERENCES:
- [Derived] Leszkowicz J, Nazar W, Wysokinska-Zakrzewska K, Zdun-Ryzewska A, Czadek-Asner P, Dettlaff-Dunowska M, Plata-Nazar K, Szlagatys-Sidorkiewicz A. Mobile app improves treatment of functional constipation in children: a randomized single-blind study. BMC Pediatr. 2025 Dec 9;25(1):980. doi: 10.1186/s12887-025-06385-y. PMID 41366315

DOCUMENTS (1):
  • Informed Consent Form (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT07025135/ICF_000.pdf